CLINICAL TRIAL: NCT05736536
Title: Health Intervention on Behaviour Change to Act for Adults With Type 2 Diabetes Mellitus and Body Mass Index of ≥ 23kg/m2: a Quasi-Experimental Study
Brief Title: Behavior Intervention for Weight Loss for Type 2 Diabetes Mellitus Adults With Obesity Problem (BMI of ≥23kg/m2)
Acronym: BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Noraini Binti Mohd Saad, Principal Investigator, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UiTMara Chance2Act
Record Dates: First submitted 2023-02-05; First posted 2023-02-21 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Behavior
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will receive a package of health education modules through Chance2Act website in addition to the existing health education being offered in the health clinic.
  Interventions: Behavioral: Chance2Act
- Control Group (No Intervention): This group will receive the existing health education being offered in the health clinic.

INTERVENTIONS:
Behavioral: Chance2Act — A Health education package that has been developed based on Transtheoretical Model to encourage behaviour change for weight loss among overweight/obese type 2 diabetes adults.
  Arms: Intervention Group

SUMMARY:
This quasi-experimental study aims to determine the effectiveness of a health intervention (Chance2Act) on behaviour change to act for weight loss among overweight/obese type 2 diabetes adults.

The main question it aims to answer is:

- Is the new health intervention (Chance2Act) effective in changing overweight/obese type 2 diabetes adults from not being ready to act, to take action to lose weight?

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients under follow-up of government health clinics Kuantan, Pahang.
* Age between 20 - 65 years old.
* Body Mass Index of more or equal to 23 kg/m2.
* In the stage of pre-contemplation, contemplation, or preparation stage of change based on the S-weights questionnaire.
* Able to understand, read and write in the Malay Language.
* Have access to smartphone devices and internet services.
* Have immediate family members (adults) who are living in the same household.

Exclusion Criteria:

* Pregnant patients.
* Patients' advanced comorbidity that will affect participation in the study protocol (e.g. vision problem, unable to walk or physically unfit to stand up, advanced heart failure, or cancer).
* Patients with mental conditions which will affect understanding of the study protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Changes of readiness to change for weight loss (behaviour) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The stage of change for weight loss is based on the S-weight questionnaire (Transtheoretical Model).
  Data type:
  Categorical data (either in pre-contemplation, contemplation, preparation, or action stage)

SECONDARY OUTCOMES:
Changes of self-efficacy for weight loss (behaviour) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes for self-efficacy to control eating impulses based on Weight Efficacy Lifestyle Questionnaire (Transtheoretical Model).
  Domains (4 items in each domain)
  * Negative emotions
  * Availability
  * Social Pressure
  * Physical discomfort
  * Positive Activities
  Data type: Numerical data. A higher score shows better outcomes. Rating of each item: 0 - 9
  Lowest score: 0 in each subscale Highest score: 36 in each subscale
Changes of decisional balance for weight loss (behaviour) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes for decisional balance to decide on the pros and cons of weight loss based on the Decisional Questionnaire Inventory questionnaire (Transtheoretical Model).
  Domains (10 items in each domain)
  * Pro scale (Measure the positive effects from weight loss. A higher score shows better outcomes)
  * Con scale (Measure the negative effects from weight loss. A higher score shows worse outcomes)
  Rating of each item: 1 - 5
  Data type: Numerical data.
  Lowest score: 10 in each subscale Highest score: 50 in each subscale
Changes in family support for healthy diet and physical activity to encourage weight loss (social support) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes for social support for weight loss based on the Social Support Scale for Diet and Exercise
  Domains:
  * Family support for physical activity (12 items)
  * Family encouragement for healthy diet (5 items)
  * Family discouragement for healthy diet (5 items)
  Rating for each item: 1 - 5
  Data type: Numerical data.
  Total subscale score:
  Family support for physical activity: 12 - 60: A higher score shows better outcomes.
  Family encouragement for healthy eating 5 - 25: A higher score shows better outcomes.
  Family discouragement for healthy eating 5 - 25: A higher score shows worse outcomes
Changes body mass index (anthropometric) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes body mass index measurement
Changes waist circumference (anthropometric) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes waist circumference measurement
Changes in body fat composition (anthropometric) | T0 (Week 0), T1 (Week 5), T2 (Week 9)
  The changes in body fat composition (total and visceral fat)

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Beserah Health Clinic, Kuantan, Pahang
  - Paya Besar Health Clinic, Kuantan, Pahang

IPD SHARING:
Plan to Share IPD: No
All data collected in the study will not be shared with other researchers to protect the confidentiality of patients' information as requested by the study site's authorized organization.
  The study IPD includes:
  1. Study Protocol
  2. Statistical Analysis Plan
  3. Informed Consent Form
  4. Clinical Study Report
  5. Analytic Code

REFERENCES:
- [Derived] Mohd Saad N, Mohamad M, Mat Ruzlin AN. Web-Based Intervention to Act for Weight Loss in Adults With Type 2 Diabetes With Obesity (Chance2Act): Protocol for a Nonrandomized Controlled Trial. JMIR Res Protoc. 2024 Jan 31;13:e48313. doi: 10.2196/48313. PMID 38294848